CLINICAL TRIAL: NCT01711502
Title: Epidemiology and Therapeutic Management of Metastatic Breast Cancer in Romania: A Retrospective Cohort Study
Brief Title: Epidemiology and Management of Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-ORO-XXX-2012/1
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Breast Cancer Nos Metastatic Recurrent
Keywords: metastatic breast cancer,; epidemiology,; retrospective cohort
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Female patients diagosed with metastatic breast cancer

SUMMARY:
This is a multicenter, national, retrospective chart-review study that will be based on the collection of data from electronical or paper-based medical records with available data on female patients diagnosed with metastatic brest cancer . The main purpose of this study is to provide accurate, evidence based description on the incidence of progression of metastatic breast cancer and its clinical management.

DETAILED DESCRIPTION:
Epidemiology and Therapeutic Management of Metastatic Breast Cancer in Romania: A retrospective cohort study

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18 years and over Diagnosis of breast cancer according to ICD-10 diagnostic criteria with confirmed metastasis
* Confirmed diagnosis between 1st July 2010 - 30th June 2011
* Female patient managed for her disease at the same setting where final diagnosis of MBC was performed

Exclusion Criteria:

* History of concurrent or other primary malignancies (except curatively resected non-melanoma skin cancer or in situ cervical cancer)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients diagosed with metastatic breast cance, age > 18 years
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The incidence rate of progression of disease in a cohort of patients newly diagnosed with MBC, either De Novo or having progressed from a non-metastatic stage | At 12 and 18 months after diagnosis

SECONDARY OUTCOMES:
The progression free survival (PFS) rates | At 12 and 18 months after diagnosis
The progression free survival (PFS) time | At 18 months after diagnosis
Time to progression (TTP) | At 18 months after diagnosis
The clinical and pathological characteristics of newly diagnosed MBC patients | At 18 months after diagnosis
The socio-demographic and anthropometric characteristics of newly diagnosed MBC patients | At 18 months after diagnosis
Health care utilization associated with the disease in Romania | At 18 months after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Dediu Mrcea, SENIOR PHYSICIAN, Principal Investigator — Bucharest Institute of Oncology; Alexandru Eniu, SENIOR PHYSICIAN, Principal Investigator — Cluj Institute of Oncology
Locations (15):
- Romania (15):
  - Doina Coste Gherasim, Baia Mare
  - Daniel Ciurescu, Brasov
  - Dana Lucia Stanculeanu, Bucharest
  - Dragos Median, Bucharest
  - Mircea Dediu, Bucharest
  - Rodica Tudor, Bucharest
  - Alexandru Eniu, Cluj-Napoca
  - Gabriela Morar Bolba, Cluj-Napoca
  - Bena Sandra, Craiova
  - Nelly Cherciu, Craiova
  - Diana Petroiu, Iași
  - Simona Angelescu, Târgovişte
  - Cristina Oprean, Timișoara
  - Stefan Curescu, Timișoara
  - Cristina Elen Pirau, Vaslui